CLINICAL TRIAL: NCT00439894
Title: Protein Phosphorylation Ancillary Study to Amgen Protocol 20060104: Open Label Study to Assess the Safety and Immunogenicity of Etanercept SFP When Administered to Subjects Diagnosed With Rheumatoid Arthritis
Brief Title: Ancillary Study to Protocol 20060104
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20060364
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; etanercept; Enbrel; Amgen
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Biospecimen Retention: None Retained — no biospecimens will be retained.

GROUPS / COHORTS (1):
- blood draw: One time blood draw
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — blood draw at baseline, week 12 and week 24

SUMMARY:
Ancillary study to the Etanercept protocol 20060104. Subjects have been asked to provide additional blood samples for further assessment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed Consent Meet all inclusion critieria outlined in Amgen Protocol 20060104

Exclusion Criteria:

* Meet exclusion criteria outlined in Amgen Protocol 20060104

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who enrolled in to Etanercept SFP 20060104 study and signed the 20060364 informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To explore the correlation between pheripheral blood cell protein phosphorylation assessemnts and rheumatoid arthritis disease activity. | week 24

SECONDARY OUTCOMES:
Explore the correlations to etanercept clinical response (ACR and DAS scores) may also be explored. | week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com